CLINICAL TRIAL: NCT03391492
Title: Invasive Pulmonary Aspergillosis Complicating Influenza Infection in Critically Ill Patients: a Prospective, Observational, Multicenter Case Control Registration Study
Brief Title: Invasive Pulmonary Aspergillosis Complicating Influenza Infection
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: Basilicum
Record Dates: First submitted 2017-12-08; First posted 2018-01-05 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Influenza With Pneumonia; Aspergillosis Invasive
Keywords: ICU

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- influenza group: All consecutive patients older than 18 years ,admitted to the ICU with respiratory distress with microbiologically confirmed diagnosis of influenza
- control group: All consecutive patients older than 18 years, admitted to the ICU for respiratory distress due to community-acquired pneumonia (CAP) and with a microbiologically confirmed absence of influenza,

SUMMARY:
Study the incidence and outcome of invasive pulmonary aspergillosis (IPA) in ICU patients with severe influenza and in influenza-negative control patients with severe community-acquired pneumonia

DETAILED DESCRIPTION:
This prospective multicentre case-control registration study in Dutch and Belgian ICUs will assess the difference in incidence and outcome of invasive pulmonary aspergillosis (IPA) in ICU patients with severe influenza compared with influenza-negative control patients with severe community-acquired pneumonia during the coming three influenza seasons (2017-2020). The study will further assess the differences in clinical characteristics and risk factors between influenza patients with and without invasive aspergillosis.

All consecutive patients aged 18 or older admitted to ICU during the inclusion period with respiratory distress due to influenza positive/negative community acquired pneumonia (CAP) will be included.

ELIGIBILITY:
Inclusion Criteria:

* patient older than 18 years,admitted to ICU with respiratory distress with microbiologically confirmed diagnosis of influenza (for inclusion in the influenza group)
* patients older than 18 years, admitted to ICU for respiratory distress due to community-acquired pneumonia , with a microbiologically confirmed absence of influenza (for inclusion in the control group)

Exclusion Criteria:

* age < 18 year
* no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients admitted from home to ICU with respiratory distress, with documented pulmonary infiltrates and initiation of antimicrobial therapy because community acquired pneumonia is the primary diagnosis or in the differential diagnosis.
  Confirmation of presence or absence of influenza is based on probe-based reverse-transcriptase polymerase chain reaction (RT-PCR) for influenza A or B directly on sputum, bronchial aspirate, broncho-alveolar (BAL) fluid or a nasopharyngeal swab.
Sampling Method: Non-Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
incidence IPA between ICU patients with severe influenza and in influenza-negative control patients | from date of admission in ICU assessed up to ICU discharge, approximately 21 days
  incidence of mycological evidence of Aspergillus and at least one Aspergillus compatible sign or symptom and radiological abnormalities based on Chest CT or Chest X ray. Mycological evidence can be provided by either (A) a positive culture of Aspergillus cultured from bronchoalveolar lavage (BAL) sample, (B) ≥2 positive cultures of Aspergillus cultured from a sputum or a bronchial aspirate or (C) a galactomannan (GM) optical density of ≥1 in BAL or ≥0.5 in serum. Aspergillus compatible signs or symptoms are defined as at least one of the following:
  * Worsening respiratory insufficiency in spite of proper antibiotic and ventilator support
  * Dyspnea
  * Haemoptysis
  * Fever refractory to at least 3 days of appropriate antibiotic (AB) therapy. Recrudescent fever after a period of defervescence of at least 48 h while still on AB without apparent cause.
  The presence of hyphae in lung biopsy or autopsy are also considered as sufficient evidence for IPA.

SECONDARY OUTCOMES:
variations in baseline factors and risk factors between influenza and non-influenza patients in ICU | from date of admission in ICU to date of ICU discharge, approximately 21 days
  difference in baseline factors: demographic, biochemical, microbiological and radiological data
rate of IPA disease progression | from date of admission to ICU to date of discharge from ICU, approximately 21 days
  rate of IPA disease progression in the subgroup of patients with IPA
rate of presence of azole resistance | from date of admission to ICU to date of discharge from ICU, approximately 21 days
  rate of presence of azole resistance in the subgroup of patients with IPA

CONTACTS AND LOCATIONS:
Overall Officials: Joost Wauters, Phd, Principal Investigator — UZ Leuven
Locations (2):
- Belgium (2):
  - AZ sint Jan, Bruges
  - Jessa AH, Hasselt

IPD SHARING:
Plan to Share IPD: Undecided